CLINICAL TRIAL: NCT05423119
Title: Investigation of Neurophysiological Substrates and Clinical Behaviour for Prognosis of Rehabilitation-induced Upper Limb Recovery After Stroke: Longitudinal Cohort Study
Brief Title: Clinical Predictors of Rehabilitation-induced Arm Recovery After Stroke: Longitudinal Cohort Study
Acronym: NeuroPro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Nicola Filippini, PHD, Psychologist, IRCCS San Camillo, Venezia, Italy
Other Study IDs: Prot. 2021.10
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: rehabilitation; upper limb; prognosis; neurophysiology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: conventional therapy — upper limb rehabilitation with and without technologies

SUMMARY:
Clinical predictors of rehabilitation-induced arm recovery after stroke are still missing since literature provides evidence mainly on the spontaneous recovery path. This longitudinal cohort study aims to identify neurophysiological and behavioural features able to predict arm recovery and how it can change according to provided rehabilitation.

DETAILED DESCRIPTION:
Rationale: evidence suggests that integrity of the Cortico-Spinal Tract (CST), valid Motor Evoked Potentials (MEPs), age and neurological status are positive prognostic features for better recovery. Concurrently, dosage of rehabilitation therapy is a key factor in promoting functional recovery. However, there are no evidence suggesting whether dose of rehabilitation also influence prediction of UL motor recovery after stroke.

Aims: to define (i) predictive features for rehabilitation-induced UL recovery and (ii) the effect of rehabilitation doses.

Methods: stroke patients will be longitudinally enrolled and assessed with Magnetic Resonance Imaging, Transcranial Magnetic Stimulation (TMS), blood sample and clinical outcome measures at the beginning (T0) of rehabilitation and after 8 weeks (T1).

ELIGIBILITY:
Inclusion Criteria:

* first ever single stroke
* unilateral cortical/subcortical stroke

Exclusion Criteria:

* other neurological disease
* psychiatric disorders
* cerebellar stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients undergoing upper limb rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Change from baseline up to 8 weeks.
  Fugl-Meyer Upper Extremity is a stroke-specific scale which assesses the upper limb motor functioning in patients with post-stroke hemiplegia. There are 3 values: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The minimum value is 0 points, which corresponds to upper limb hemiplegia. The maximum value is 66 points, which corresponds to normal motor performance.

SECONDARY OUTCOMES:
Action Research Arm Test | Change from baseline up to 8 weeks.
  ARAT is a stroke-specific scale which assesses the upper limb motor activities. The maximum value is 57 and corresponds to normal motor performance
Reaching Performance Scale | Change from baseline up to 8 weeks.
  Reaching Performance Scale assesses the ability of subjects to reach an object (a cone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength. The minimum value is 0 points, which corresponds to incapacity of any ability of reaching an object. The maximum value is 36 points, which corresponds to the preservation of the ability of reaching an object.
Box & Blocks Test | Change from baseline up to 8 weeks.
  The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.
Medical Research Council | Change from baseline up to 8 weeks.
  The scale assess motor strength for each muscle tested. The score goes from 0 (no muscle contraction) to 5 (normal muscle strength against high resistance).
Imaging data | Change from baseline up to 8 weeks.
  functional and structural connectivity of the brain
Presence of Motor Evoked Potentials | Change from baseline up to 8 weeks.
  Presence of Motor Evoked Potentials in the upper limb
Modified Ashworth Scale | Change from baseline up to 8 weeks
  Spasticity is measured using the Modified Ashworth Scale of five muscles: Pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus (Total score = 20 points). The therapist evaluates the spasticity of each muscles. There are 5 values: 0 (no increase in muscle tone), 1 (slight increase in muscle tone), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone), 4 (affected part rigid in flexion or extension).
Functional Independence Measure | Change from baseline up to 8 weeks
  Functional Independence Measure scale is an 18-item scale that assesses the degree of independence in carrying out activities of daily living. There are 7 values: 1 (Total Assistance or not Testable), 2 (Maximal Assistance), 3 (Moderate Assistance), 4 (Minimal Assistance), 5 (Supervision), 6 (Modified Independence), 7 (Complete Independence). The minimum values is 18 points, which corresponds to the lower level of independence in activities of daily living. The maximum value is 126 points, which corresponds to the maximum level of independence in activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Filippiin, Principal Investigator — IRCCS San Camillo, Venezia, Italy
Locations (1):
- IRCCSSanCamillo, Lido, Venezia, Italy